CLINICAL TRIAL: NCT06984146
Title: Flat-dose Nivolumab (40 mg) in Combination With Doxorubicin, Vinblastine, and Dacarbazine (AVD) for Newly Diagnosed Advanced Classic Hodgkin Lymphoma
Brief Title: Nivo40-AVD for Advanced Classic Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nivo40-AVD
Record Dates: First submitted 2025-05-02; First posted 2025-05-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivo40-AVD (Experimental): Nivolumab 40 mg IV day 1 and 15; Doxorubicin 25 mg/m2 IV day 1 and 15; Vinblastine 6 mg/m2 IV day 1 and 15; Dacarbazine 375 mg/m2 day 1 and 15
  Interventions: Drug: Nivolumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Nivolumab — 40 mg day 1 and 15
Drug: Doxorubicin — 25 mg/m2 day 1 and 15
Drug: Vinblastine — 6 mg/m2 (not exceeding 10 mg) day 1 and 15
Drug: Dacarbazine — 375 mg/m2 day 1 and 15

SUMMARY:
The aim of the current trial is to evaluate the efficacy and safety of flat-dose nivolumab (40 mg) in combination with AVD in the management of patients with newly diagnosed advanced classic Hodgkin Lymphoma

DETAILED DESCRIPTION:
Patients will receive 6 cycles of Nivo40-AVD with interim and EOT PET/CT scan. Interim PET/CT will not affect clinical decisions and is done as part of the study on response predictors after first line PD-1 inhibitor therapy. In patients achieving only partial metabolic response after 6 cycles (Deauville score ≥ 4) radiation therapy is allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Newly-diagnosed histologically verified advanced stage (IIB-IV as per GHSG) classic Hodgkin lymphoma
2. No past history of autoimmune disease
3. Age > 18 years
4. Ejection fraction > 50%
5. ECOG 0-4

Exclusion Criteria:

1. Organ failure (e.g. creatinine > 2x ULN; ALT or AST > 5x ULN; bilirubin > 2x ULN; hemodynamic instability; respiratory failure > Grade 1)
2. Uncontrolled infection
3. Pregnancy
4. Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Complete remission and complete metabolic response | 2 years
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Kaprin, Study Chair — FSBI "National Medical Research Radiological Centre" (NMRRC) of the Ministry of Health of the Russian Federation
Locations (1):
- P. Hertsen Moscow Oncology Research Institute (MORI) for administrative and economic work - the branch of the FSBI "National Medical Research Radiological Centre" (NMRRC) of the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data might not be shared to protect patient privacy and confidentiality. All other information regarding the study will be published in detail